CLINICAL TRIAL: NCT01261910
Title: Enhancing Education Regarding Living Donor Transplant Among Kidney Transplant Candidates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Barnabas Medical Center (Other)
Collaborators: University of Medicine and Dentistry of New Jersey (Other); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SBMC-2009-53
Record Dates: First submitted 2010-12-14; First posted 2010-12-17 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Kidney Transplant; Living-Donor Kidney Transplant; Chronic Kidney Disease; End-stage Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual education (standard care) (No Intervention): On the day of the transplant evaluation at the transplant center, participants receive usual transplant education regarding living donor kidney transplant.
- Intensive initial education (Experimental): On the day of the transplant evaluation at the transplant center, participants receive usual transplant education regarding living donor kidney transplant. In addition, participants will (1) view a video, brochure, and fact sheet regarding living kidney donation, and (2) discuss the videos and materials with a transplant educator, in-person.
  Interventions: Behavioral: Intensive initial education

INTERVENTIONS:
Behavioral: Intensive initial education — Participants will (1) view a video, brochure, and fact sheet regarding living kidney donation, and (2) discuss the videos and materials with a transplant educator, in-person.
  Arms: Intensive initial education

SUMMARY:
The primary purpose of this study is to test different methods by which kidney transplant centers can educate potential transplant candidates about living donor kidney transplant (LDKT).

The most effective ways to educate kidney transplant candidates about LDKT remain unclear. The goal is to determine, among a diverse cohort of potential kidney transplant candidates, whether a transplant center-based intervention will increase understanding of the opportunities for and process, risks, and benefits of living kidney donation and LDKT. The investigators hypothesize that kidney transplant candidates' understanding of living kidney donation and LDKT will be increased by interventions implemented at the transplant center on the day of transplant evaluation.

The investigators propose a single-center, 2-arm, cluster-randomized, controlled trial to compare the effects of two educational strategies upon transplant candidates' understanding of living kidney donation and LDKT:

1. Usual transplant education implemented by the transplant center, on the day of the transplant evaluation (standard care); and
2. Intensive initial transplant education implemented on the day of the transplant evaluation.

Intensive initial transplant education will utilize videos of living donors' experiences as well as a session with a trained Transplant Educator, who will focus upon living donation education. One week after the transplant evaluation day and 3 months later, the investigators will assess transplant candidates' knowledge of LDKT (using questionnaires), identify correlates of increased understanding of LDKT, and assess racial/ethnic differences in the understanding of LDKT.

ELIGIBILITY:
Inclusion Criteria:

* Appear for initial kidney transplant evaluation at Saint Barnabas Medical Center
* 18 years of age or older
* Able to provide informed consent
* Able to speak, hear, and understand English

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2010-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Knowledge and understanding of the opportunities for and process, risks, and benefits of living kidney donation and LDKT | Up to 1 week after the transplant education day

SECONDARY OUTCOMES:
Knowledge and understanding of the opportunities for and process, risks, and benefits of living kidney donation and LDKT | Three months after the transplant education day
Attitudes, confidence, and opinions regarding living kidney donation and LDKT | (1) Up to 1 week after the transplant education day, and (2) Three months after the transplant education day
Changes in knowledge/understanding and attitudes/confidence/opinions regarding living kidney donation and LDKT | (1) Up to 1 week after the transplant education day, and (2) Three months after the transplant education day, compared to prior to the transplant evaluation day (baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Francis L Weng, MD, Principal Investigator — St. Barnabas Medical Center
Locations (1):
- Saint Barnabas Medical Center, Livingston, New Jersey, United States

REFERENCES:
- [Derived] Campbell ZC, Dawson JK, Kirkendall SM, McCaffery KJ, Jansen J, Campbell KL, Lee VW, Webster AC. Interventions for improving health literacy in people with chronic kidney disease. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD012026. doi: 10.1002/14651858.CD012026.pub2. PMID 36472416
- [Derived] Weng FL, Brown DR, Peipert JD, Holland B, Waterman AD. Protocol of a cluster randomized trial of an educational intervention to increase knowledge of living donor kidney transplant among potential transplant candidates. BMC Nephrol. 2013 Nov 19;14:256. doi: 10.1186/1471-2369-14-256. PMID 24245948